CLINICAL TRIAL: NCT01595113
Title: A Follow-up Observational Study of Safety of Clinical Trial Conducted With Cell Transplant Therapy Using Hearticellgram-AMI for Patients With Acute Myocardial Infarction
Brief Title: Safety Study of Clinical Cell Transplant Therapy Using Hearticellgram-AMI for Patients With Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PMC-BD-CT-P-001
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2013-11

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the safety of the previously conducted clinical trial cell transplant therapy using Hearticellgram-AMI for patients with acute myocardial infarction. This is a follow-up observational study and targeting the subjects who participated in the previously conducted clinical trial.

DETAILED DESCRIPTION:
The safety evaluation in this clinical trial is performed with variables, such as occurrence and severity of adverse events, clinical laboratory tests, vital signs, physical examination, cardiac events, and cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have elapsed for more than 2 years after onset of acute myocardial infarction among the patients who had received cell transplant therapy or drug treatment at least once in test and control group on the previously conducted clinical trial.
* Subjects agreed to participate in this follow-up study and signed the consent form.

Exclusion Criteria:

* N/A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects agreed to participate in this follow-up observational study among the subjects (80 patients:40-test group, 40-control group) who participated in the previously conducted clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Soo Ahn, Principal Investigator — Wonju Severance Christian Hospital